CLINICAL TRIAL: NCT02216786
Title: A Randomized Phase II Study of Fulvestrant in Combination With the Dual mTOR Inhibitor AZD2014 or Everolimus or Fulvestrant Alone in Estrogen Receptor-positive Advanced or Metastatic Breast Cancer
Brief Title: A Randomized Study of AZD2014 in Combination With Fulvestrant in Metastatic or Advanced Breast Cancer
Acronym: MANTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 009175QM
Record Dates: First submitted 2014-03-12; First posted 2014-08-15 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Estrogen Receptor Positive Breast Cancer
MeSH Terms: interventions — vistusertib; Everolimus; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fulvestrant and AZD2014 (continuous) (Experimental): Experimental arm
  Interventions: Drug: AZD2014; Drug: Fulvestrant
- Everolimus and Fulvestrant (Active Comparator): Comparator arm
  Interventions: Drug: Everolimus; Drug: Fulvestrant
- Fulvestrant (Active Comparator): Control 1
  Interventions: Drug: Fulvestrant
- Fulvestrant +AZD2014 (intermittent) (Experimental): Experimental arm
  Interventions: Drug: AZD2014; Drug: Fulvestrant

INTERVENTIONS:
Drug: AZD2014 — Oral tablet
  Arms: Fulvestrant +AZD2014 (intermittent); Fulvestrant and AZD2014 (continuous)
Drug: Everolimus — Oral tablet
  Other Names: Afinitor
  Arms: Everolimus and Fulvestrant
Drug: Fulvestrant — Im injection
  Other Names: Faslodex

SUMMARY:
This is an open-label, multicentre, 4-arm randomised phase II trial of fulvestrant + AZD2014 versus fulvestrant + everolimus versus fulvestrant alone in patients with ER-positive, HER2-negative advanced or metastatic breast cancer, whose disease relapsed during treatment with (or within 12 months after discontinuation of) an AI in the adjuvant setting or progressed during treatment with an AI in the metastatic setting. Patients will be randomised (2:3:3:2) to one of the four treatment arms:

* Fulvestrant
* Fulvestrant + AZD2014 (continuous daily schedule)
* Fulvestrant + AZD2014 (intermittent schedule - 2 days on, 5 days off)
* Fulvestrant + everolimus

Randomization will be stratified by the following criteria:

* Measurable disease (vs. non-measurable).
* Sensitivity to prior endocrine therapy (sensitive versus resistant)

DETAILED DESCRIPTION:
This is an open-label, multicentre, 4-arm randomised phase II trial of fulvestrant + AZD2014 versus fulvestrant + everolimus versus fulvestrant alone in patients with ER-positive, HER2-negative advanced or metastatic breast cancer, whose disease relapsed during treatment with (or within 12 months after discontinuation of) an AI in the adjuvant setting or progressed during treatment with an AI in the metastatic setting. Patients will be randomised (2:3:3:2) to one of the four treatment arms:

* Fulvestrant
* Fulvestrant + AZD2014 (continuous daily schedule)
* Fulvestrant + AZD2014 (intermittent schedule - 2 days on, 5 days off)
* Fulvestrant + everolimus

Randomization will be stratified by the following criteria:

* Measurable disease (vs. non-measurable).
* Sensitivity to prior endocrine therapy (sensitive versus resistant) Sensitivity to prior endocrine therapy is defined as (i) at least 24 months of endocrine therapy before recurrence in the adjuvant setting or (ii) a complete or partial response to prior metastatic endocrine treatment, or (iii) stabilization for at least 24 weeks of endocrine therapy for advanced disease.

Treatment will be continued until disease progression unless there is evidence of unacceptable toxicity or if the patient requests to be withdrawn from the study. If one of the treatments (fulvestrant or mTOR inhibitor) is discontinued prior to disease progression, patients should be continued on single agent treatment until progression, evidence of unacceptable toxicity or if the patient requests to be withdrawn from the study.

At the time of documented disease progression (using RECIST 1.1), patients randomised to receive fulvestrant + everolimus who still meet eligibility criteria may be permitted to receive open-label crossover treatment with fulvestrant + AZD2014. Crossover therapy must begin no later than 28 days after the clinic visit at which progression was determined. Patients will receive crossover therapy until progression, intolerable toxicity, elective withdrawal from the study, or until the completion or termination of the study, whichever occurs first.

Tumour evaluations will be performed before the initiation of treatment, every 8 weeks during the first 40 weeks and every 12 weeks thereafter until disease progression.

The study will also assess the relationship between the anticipated anti-tumour activity of the treatment regimen and biological characteristics of patients' tumour at baseline

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent prior to admission to this study
2. Women, age ≥18 years
3. Histologically confirmed breast cancer
4. Metastatic or locally recurrent disease; locally recurrent disease must not be amenable to resection with curative intent (patients who are considered suitable for surgical or ablative techniques following potential down-staging with study treatment are not eligible).
5. Patients must have:

   1. at least one lesion, not previously irradiated, that can be measured accurately at baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have short axis ≥ 15mm) with computed tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements, or
   2. lytic or mixed (lytic + sclerotic) bone lesions in the absence of measurable disease as defined above; patients with sclerotic/osteoblastic bone lesions only in the absence of measurable disease are not eligible
6. Radiological or clinical evidence of recurrence or progression
7. ER-positive disease
8. HER2-negative disease with 0, 1+ or 2+ intensity on IHC and no evidence of amplification on ISH.
9. Formalin fixed, paraffin embedded tumour sample from the primary and/or recurrent cancer must be available for central testing
10. Postmenopausal women.
11. Disease refractory to aromatase inhibitors (AI)
12. Haematologic and biochemical indices within acceptable limits
13. ECOG performance status 0-2
14. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had a hysterectomy, bilateral oophorectomy, bilateral tubular ligation or is post-menopausal (total cessation of menses for ≥ 1 year

Exclusion criteria:

1. Presence of life-threatening metastatic visceral disease, defined as extensive hepatic involvement or any degree of brain or leptomeningeal involvement (past or present), or symptomatic pulmonary lymphangitic spread. Patients with discrete pulmonary parenchymal metastases are eligible, provided their respiratory function is not compromised as a result of disease.
2. More than one line of prior chemotherapy for metastatic breast cancer
3. Prior chemotherapy, biological therapy, androgens, thalidomide, immunotherapy, other anticancer agents or any investigational agents within 14 days of starting study treatment (not including palliative radiotherapy at focal sites), radiotherapy with a wide field of radiation (greater than or equal to 30% marrow or whole pelvis or spine) within 4 weeks of starting study treatment, or strontium-90 (or other radiopharmaceuticals) within the past 3 months or major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access); with the exception of alopecia, all unresolved toxicities from prior treatment should be no greater than CTCAE grade 1 at the time of starting study treatment
4. Prior treatment with fulvestrant or everolimus
5. Prior treatment with PI3K inhibitors, Akt inhibitors or other mTOR inhibitors.
6. Patients receiving concomitant immunosuppressive agents or chronic systemic corticosteroids (≥10 mg prednisolone or an equivalent dose of other anti-inflammatory corticosteroids) use for ≥28 days at the time of study entry except in cases outlined below: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed. Patients on stable low dose of corticosteroids for at least two weeks before randomisation are allowed
7. Current refractory nausea and vomiting, chronic gastrointestinal disease or inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of the study medication
8. Clinically significant pulmonary dysfunction
9. Significant cardiovascular disease
10. QTc prolongation defined as a QTc interval >470 msecs or other significant ECG abnormalities including 2nd degree (type II) or 3rd degree AV block or bradycardia (ventricular rate <50 beats/min)
11. Concomitant medications known to prolong QT interval, or with factors that increase the risk of QTc prolongation or risk of arrhythmic events (such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age)
12. Clinically significant abnormalities of glucose metabolism
13. Exposure to potent or moderate inhibitors or inducers of CYP3A4/5 within 2 weeks before the first dose of study treatment
14. Exposure to potent or moderate inhibitors or inducers of CYP2C8 within 1 week before the first dose of study treatment.
15. Application of haemopoietic growth factors (e.g. G-CSF, GM-CSF) within 2 weeks before receiving study drug
16. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
17. History of hypersensitivity to active or inactive excipients of AZD2014 or everolimus or drugs with a similar chemical structure or class to AZD2014 or everolimus
18. History of hypersensitivity to active or inactive excipients of fulvestrant and/or castor oil.
19. Patients presenting with anaemia symptoms (haemoglobin ≤ 90 g/L).
20. Currently receiving (and are unwilling to discontinue) oestrogen replacement therapy (last dose ≤ 7 days prior to randomisation)
21. Psychological, familial, sociological or geographical conditions that do not permit compliance with the study protocol.
22. Detained persons or prisoners
23. Pregnant or nursing women (including no breast feeding from two weeks before the first dose of study medication, till 8 weeks after the last dose of study medication).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2014-01-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Date of randomisation to date of first documented progression, assessed up to 100 weeks
  Defined as the time from the date of randomisation to the date of first documented tumour progression based on investigator assessment (using RECIST 1.1) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free survival | time from the date of randomisation to the date of first documented tumour progression, assessed up to 100 weeks
  Progression-free survival, defined as the time from the date of randomisation to the date of first documented tumour progression as assessed by an independent review facility [IRF] (using RECIST 1.1) or death from any cause, whichever occurs first.
Objective response | Time from date of randomisation to documented objective response, assessed up to 60 months
  Time from date of randomisation to documented objective response, defined as a complete or partial response, based on investigator and IRF assessment (using RECIST 1.1)
Average change (%) in tumour size | 16 weeks after baseline
  Average change (%) in tumour size at 16 weeks compared to baseline, based on investigator and IRF assessment using RECIST 1.1; tumour size is defined as the sum of the longest diameters of the target (i.e. measurable tumour) lesions
Clinical Benefit (CB) | Date of randomisation to 24 weeks.
  Clinical Benefit (CB), defined as number of patients with complete or partial response or stable disease maintained ≥24 weeks, based on investigator and IRF assessment using RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, Prof, Principal Investigator — Queen Mary's University of London
Locations (79):
- France (5):
  - ICO Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Antoine Lacassagne Centre De Lutte Contre Le Cancer De Nice, Nice
  - Hospital Center Private Saint-Grégoire, Saint-Grégoire
  - Centre Paul Strauss, Strasbourg
- Georgia (4):
  - Clinic Health House, Tbilisi
  - Institute of Clinical Oncology, Tbilisi
  - S. Khechinashvili University Clinic, Tbilisi
  - Tbilisi Cancer Center, Tbilisi
- Germany (15):
  - Frauenärztliche Gemeinschaftspraxis - Onkologie, Braunschweig
  - Kliniken Essen-Mitte Senologie, Essen
  - Klinik für Gynäkologie & Geburtshilfe/Brustzentrum, Frankfurt
  - Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau
  - MediProjekt GbR Hannover, Hannover
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Dokusan GmbH, Herne
  - St. Vincentius Kliniken, Karlsruhe
  - Schwerpunktpraxis Hämatologie / Onkologie MVZ Lahr, Lahr
  - Klinikum Neumarkt, Neumarkt
  - Onkologische Praxis, Oldenburg
  - Praxis für Innere Medizin, Singen
  - MVZ Klinik Dr. Hancken GmbH, Stade
  - Mutterhaus der Borromäerinnen, Trier
  - Schwarzwald Baar Klinikum, Villingen-Schwenningen, Villingen-Schwenningen
- Hungary (4):
  - Uzsoki Street Hospital, Budapest
  - Bacs-Kiskun County Hospital, Kalocsa
  - University of Pecs, Institute of Oncology, Pécs
  - Zala County Szent Rafael Hospital, Zalaegerszeg
- Portugal (2):
  - Hospital da Luz, Lisbon
  - Ipo Porto, Porto
- Romania (5):
  - Center of Oncology Euroclinic, Bucharest
  - Oncology Center Sf Nectarie, Caracal
  - Cluj County Clinical Emergency Hospital, Clinical Department of Medical Oncology, Cluj-Napoca
  - Oncology Institute "Prof. Dr. Ion Chiricuta", Cluj-Napoca
  - Oncology Center Oncolab Craiova, Craiova
- South Korea (3):
  - National Cancer Center South Korea, Goyang
  - Korea University Medical Center Guro Hospital, Seoul
  - Yonsei University Health System, Seoul
- Spain (11):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Instituto Oncologico Dr. Rosell, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castelló
  - Cafeteria Hospital San Pedro de Alcantara, Cáceres
  - Hospital Ico Josep Trueta, Girona
  - University Hospital Arnau de Vilanova, Lleida
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Son Llàtzer, Palma
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitari Sant Joan de Reus, Tarragona
- United Kingdom (30):
  - Wansbeck General Hospital, Ashington
  - Princess of Wales Hospital, Bridgend
  - Royal Sussex County Hospital, Brighton
  - Kent and Canterbury Hospital, Canterbury
  - Cumberland Infirmary, Carlisle
  - Broomfield Hospital, Chelmsford
  - University Hospital of North Durham, Durham
  - Calderdale Royal Hospital, Halifax
  - Huddersfield Royal Infirmary, Huddersfield
  - Kidderminster Hospital, Kidderminster
  - Royal Glamorgan Hospital, Llantrisant
  - Queen Mary University of London, London
  - Charring Cross Hospital, London
  - King's College Hospital, London
  - Mount Vernon Hospital, London
  - Queen Elizabeth Hospital, Woolwich, London
  - Saint Bartholomew's Hospital, London
  - The Royal Free Hospital, London
  - The Kent Oncology Centre, Maidstone
  - North Tyneside General Hospital, North Shields
  - Nottingham City Hospital, Nottingham
  - Derriford Hospital, Plymouth
  - Weston Park Hospital, Sheffield
  - Solihull Hospital, Solihull
  - Southend University Hospital, Southend-on-Sea
  - Royal Stoke University Hospital, Stoke-on-Trent
  - King's Mill Hospital, Sutton in Ashfield
  - Great Western Hospital, Swindon
  - Wrexham Maelor, Wrexham
  - Yeovil District Hospital, Yeovil

REFERENCES:
- [Result] Schmid P, Zaiss M, Harper-Wynne C, Ferreira M, Dubey S, Chan S, Makris A, Nemsadze G, Brunt AM, Kuemmel S, Ruiz I, Perello A, Kendall A, Brown J, Kristeleit H, Conibear J, Saura C, Grenier J, Mahr K, Schenker M, Sohn J, Lee KS, Shepherd CJ, Oelmann E, Sarker SJ, Prendergast A, Marosics P, Moosa A, Lawrence C, Coetzee C, Mousa K, Cortes J. Fulvestrant Plus Vistusertib vs Fulvestrant Plus Everolimus vs Fulvestrant Alone for Women With Hormone Receptor-Positive Metastatic Breast Cancer: The MANTA Phase 2 Randomized Clinical Trial. JAMA Oncol. 2019 Nov 1;5(11):1556-1564. doi: 10.1001/jamaoncol.2019.2526. PMID 31465093